CLINICAL TRIAL: NCT00438802
Title: A Phase I Study of Alefacept (AmeviveTM) in the Treatment of Cutaneous T-cell Lymphoma and Peripheral T-cell NHL
Brief Title: Alefacept in Treating Patients With Relapsed or Refractory Cutaneous T-Cell Lymphoma or Peripheral T-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000530071; P50CA097274 (NIH); P30CA015083 (NIH); LS058C (Other: Mayo Clinic Cancer Center); 06-002246 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2016-03

CONDITIONS: Lymphoma
Keywords: recurrent cutaneous T-cell non-Hodgkin lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; adult nasal type extranodal NK/T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Extranodal NK-T-Cell; Mycosis Fungoides; Sezary Syndrome | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- alefacept (Experimental): Determine both the maximum tolerated dose level as well as the optimal immunologic dose and toxicity.
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — Dose escalation theme. 0.075mg/kg by IV Weekly x 8 to 0.30mg/kg IV Weekly x 8
  Other Names: Amevive

SUMMARY:
RATIONALE: Combinations of biological substances in alefacept may be able to carry cancer-killing substances directly to cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of alefacept in treating patients with relapsed or refractory cutaneous T-cell lymphoma or peripheral T-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose or the optimal immunologic dose of alefacept in patients with relapsed or refractory cutaneous T-cell lymphoma or peripheral T-cell non-Hodgkin's lymphoma.

Secondary

* Determine if antitumor activity of this drug exists in these patients.

OUTLINE: This is a multicenter, dose-escalation study.

* Induction therapy: Patients receive alefacept IV over 2-5 minutes once weekly for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable disease or complete or partial response after induction therapy proceed to maintenance therapy.

Cohorts of 6 patients receive escalating doses of alefacept until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. The optimal immunologic dose is defined as the dose that does not exceed the MTD, has the highest alefacept level, and achieves saturation of CD2 receptors.

* Maintenance therapy: Patients receive alefacept IV on day 1. Treatment repeats every 4 weeks for 10-12 courses in the absence of disease progression or unacceptable toxicity.

Patients who experience disease progression during maintenance therapy may receive reinduction therapy* comprising 4 weekly doses of alefacept. The patient then proceeds to a second maintenance phase in the absence of disease progression.

NOTE: *Only 1 reinduction allowed.

Patients undergo blood and tissue collection periodically for pharmacological studies. Blood serum is analyzed for alefacept concentration, cytokine concentration, CD16 polymorphisms, and CD2 saturation via flow cytometry.

After completion of study treatment, patients are followed every 3 months for up to 3 years and then periodically thereafter.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell lymphoma (CTCL) or peripheral T-cell non-Hodgkin's lymphoma

  * Diagnostic biopsies must have been obtained within the past 6 months
* Relapsed or refractory disease

  * Patients with CTCL must have failed ≥ 2 skin-directed therapies

    * No limit on the number of prior therapies
* Measurable disease, defined as at least 1 bidimensionally measurable lesion > 2 cm by CT scan, MRI, physical exam, or photograph with appended ruler

  * At least 2 bidimensionally measurable target lesions required for patients with skin lesions only
* No CNS lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 2 times upper limit of normal (ULN) OR direct bilirubin ≤ 1.5 times ULN
* AST ≤ 3 times ULN (≤ 5 times ULN if liver involvement)
* Creatinine ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to provide all research blood samples as required by the protocol
* Willing to undergo repeat biopsy of either an accessible skin lesion or lymph node, if there are no circulating sezary cells, for the purpose of research studies (patients without easily accessible lesions are not required to have a repeat biopsy solely for research purposes but must be willing to provide a portion of the on-study biopsy or a previous lymphoma biopsy, if available)
* No known congenital or acquired immunodeficiency syndromes, including HIV
* No known active viral hepatitis or tuberculosis infection
* No uncontrolled infection
* No other uncontrolled serious medical condition unrelated to lymphoma (e.g., cardiac arrhythmia or diabetes)
* No other active malignancies
* No history of serious allergic reaction to citrate or glycine

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior cytotoxic chemotherapy
* More than 3 weeks since prior denileukin diftitox
* More than 3 weeks since prior radiotherapy (less than 3 weeks if the acute side effects of this therapy are resolved)
* More than 2 weeks since prior oral corticosteroids (unless being used to treat adrenal insufficiency)
* More than 2 weeks since prior phototherapy, including ultraviolet B and psoralen with ultraviolet A
* More than 1 week since prior biologic therapy
* No concurrent chemotherapy, other immunotherapy, or radiotherapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2010-08-24 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Starting Dose Level 1= 0.15 mg/kg> Each cycle is 4 weeks.> > Cycle 1 and 2:> Alefacept by IV Weekly>
  > Cycles 3-12:> Alefacept by IV 1 x every 4 weeks
- Dose Level 2: Starting Dose Level 1= 0.20 mg/kg> Each cycle is 4 weeks.> > Cycle 1 and 2:> Alefacept by IV Weekly>
  > Cycles 3-12:> Alefacept by IV 1 x every 4 weeks
- Dose Level 3: Starting Dose Level 1= 0.30 mg/kg> Each cycle is 4 weeks.> > Cycle 1 and 2:> Alefacept by IV Weekly>
  > Cycles 3-12:> Alefacept by IV 1 x every 4 weeks
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 6 | 8 | 9
Completed | 6 | 8 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 2: Dose Level 2= 0.20 mg/kg> Each cycle is 4 weeks.> > Cycle 1 and 2:> Alefacept by IV Weekly>
  > Cycles 3-12:> Alefacept by IV 1 x every 4 weeks
- Dose Level 3: Dose Level 3= 0.30 mg/kg> Each cycle is 4 weeks.> > Cycle 1 and 2:> Alefacept by IV Weekly>
  > Cycles 3-12:> Alefacept by IV 1 x every 4 weeks
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 6 | 8 | 9 | 23
Age, Continuous [Median (Full Range); unit: years] | 50.5 [46 to 80] | 69 [48 to 80] | 66 [56 to 76] | 64 [46 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 12
  Male | 2 | 3 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: The Maximum Tolerated Dose (MTD) will be defined as the highest safely-tolerated dose where at most one out of six patients experiences a Dose Limiting Toxicity (DLT) with the next higher dose level having at least 2 patients who have experienced DLT. The MTD determination will be based on toxicities encountered during the first 8 weeks of treatment.>
  > For this protocol, dose-limiting toxicity (DLT) will be defined as an adverse event attributed (definitely, probably, or possibly) to the study treatment and meeting the following criteria:>
  * grade 4 toxicity for neutrophils (<0.5 x 109/L) or platelets (<25 x 109/L)>
  * any grade 3 or higher solid organ toxicity not explainable by another obvious cause.>
  * more than 10 x ULN AST toxicity for more than 14 days>
  * any grade 4 infection.>
  The number of patients who reported a dose limiting toxicity is reported here.
Time Frame: 8 weeks from registration
Population: Two patients from Dose level 2 were not able to complete cycle 1 and were not evaluated for dose limiting toxicity.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Dose Level 1= 0.15 mg/kg> Each cycle is 4 weeks.> > Cycle 1 and 2:> Alefacept by IV Weekly>
  > Cycles 3-12:> Alefacept by IV 1 x every 4 weeks
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 6 | 6 | 9
Participants | 0 | 1 | 1

2. Secondary Outcome: Clinical Response
Description: Treatment response and evaluation will be performed using standardized lymphoma International Working Group recommendations.>
  > A Complete Response (CR) requires:>
  * Complete disappearance of all detectable clinical and radiographic evidence of> disease.>
  * All lymph nodes and nodal masses must have regressed to normal size.>
  Partial Response (PR):>
  * greater than 50% decrease in Sum of Product Dimensions of the six largest dominant nodes, nodal masses, or skin lesions.>
  * No increase in size of other nodes>
  * no new sites of disease.
Time Frame: up to 12 cycles (28 days per cycle) of treatment.
Population: Two patients from Dose level 2 were not able to complete cycle 1 and were not evaluated for dose limiting toxicity.
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 6 | 6 | 9
participants
  Complete Response (CR) | 1 | 0 | 0
  Partial Response (PR) | 2 | 1 | 0

3. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The Maximum Tolerated Dose (MTD) will be defined as the highest safely-tolerated dose where at most one out of six patients experiences a Dose Limiting Toxicity (DLT) with the next higher dose level having at least 2 patients who have experienced DLT. The MTD determination will be based on DLT toxicities encountered during the first 8 weeks of treatment reported in Primary Outcome Measure #1.
Time Frame: 8 weeks from registration
Population: Two patients from Dose level 2 were not able to complete cycle 1 and were not evaluated for dose limiting toxicity.
Measure: Number; unit: mg/kg Alefacept
Groups:
- All Patients: Dose Level 1= 0.15 mg/kg> Dose Level 2= 0.20 mg/kg> Dose Level 3= 0.30 mg/kg> Each cycle is 4 weeks.> > Cycle 1 and 2:> Alefacept by IV Weekly>
  > Cycles 3-12:> Alefacept by IV 1 x every 4 weeks
Arm/Group | All Patients
Number analyzed (Participants) | 21
mg/kg Alefacept | 0.30

ADVERSE EVENTS:
Groups:
- Dose Level 1; Dose Level 2; Dose Level 3: Alefacept by IV 1 x every 4 weeks
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/8 | 2/9
Other Adverse Events (participants affected / at risk) | 5/6 | 7/8 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=8) | Dose Level 3 (N=9)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=8) | Dose Level 3 (N=9)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (21) | 5 (30) | 5 (13)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (4) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Upper respiratory infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (10) | 4 (8) | 0 (0)
Leukocyte count decreased (Investigations) | 2 (6) | 1 (1) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (8) | 2 (3) | 1 (1)
Platelet count decreased (Investigations) | 2 (7) | 2 (2) | 3 (5)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (21) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes